CLINICAL TRIAL: NCT02664103
Title: A Phase II Open-label Randomized Study of a Fixed-dose Combination of Capecitabine and Cyclophosphamide Administered at Different Doses/Regimens With Metronomic Schedule in Patients With Metastatic Breast Cancer
Brief Title: Study of Capecitabine and Cyclophosphamide Administered as a Single Pill in Patients With Advanced Breast Cancer
Acronym: METRO-ABC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPCYR07568; U1111-1166-1149 (Other: UTN)
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SAR439281(Cohort 1) (Experimental): Regimen 1: one full-dose tablet containing capecitabine and cyclophosphamide, given BID without interruption
  Interventions: Drug: Fixed-dose combination of capecitabine and cyclophosphamide SAR439281
- SAR439281(Cohort 2) (Experimental): Regimen 2: two tablets containing capecitabine and cyclophosphamide, given OD without interruption
  Interventions: Drug: Fixed-dose combination of capecitabine and cyclophosphamide SAR439281
- SAR439281(Cohort 3) (Experimental): Regimen 3: one tablet containing capecitabine and cyclophosphamide, given OD without interruption
  Interventions: Drug: Fixed-dose combination of capecitabine and cyclophosphamide SAR439281

INTERVENTIONS:
Drug: Fixed-dose combination of capecitabine and cyclophosphamide SAR439281 — Pharmaceutical form:Tablet Route of administration: Oral

SUMMARY:
Primary Objectives:

* To assess the safety for each cohort of patients on a fixed-dose combination pill of capecitabine and cyclophosphamide administered at flat dose and with metronomic schedule (defined as continuous daily treatment without interruption) in patients with metastatic breast cancer.
* To assess the pharmacokinetics (PKs) and bioavailability of the fixed-dose combination pill of capecitabine and cyclophosphamide administered at different doses/regimens by metronomic schedule in patients with metastatic breast cancer.

Secondary Objectives:

* To assess antitumor activity of the fixed-dose combination pill of capecitabine and cyclophosphamide administered at different doses/regimens by metronomic schedule in patients with metastatic breast cancer given at 3 different doses and schedules (regimen 1=standard dose twice daily [BID], regimen 2=full dose once daily [OD], regimen 3=low dose [OD])
* Disease Control Rate (DCR)
* Overall Response Rate (ORR)
* Time to Progression (TTP) using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria (version 1.1).
* To evaluate the compliance under treatment.
* To describe evolution of toxicities.
* To assess safety all along patient's treatment.

DETAILED DESCRIPTION:
Primary objective will be evaluated at 12 weeks. Patients who show evidence of efficacy will be treated and followed-up until progression of the disease.

ELIGIBILITY:
Inclusion criteria:

* Female ≥18 and ≤65 years old.
* Patients with histologically or cytologically confirmed Metastatic Breast Cancer (HER2 negative, ER/PR positive or negative), who are candidates to receive capecitabine and cyclophosphamide as per Investigator's judgment, and meet either one of the following characteristics:
* Recurrence of the disease following at least 2 lines of chemotherapy failure for metastatic triple negative breast cancer.
* In ER/PR positive breast cancer, recurrence of the disease following at least 1 line of chemotherapy failure and 2 lines of hormonal therapy failure.
* Patients who have been previously treated with capecitabine can be recruited in the study provided:
* As per the Investigator's opinion, patients will benefit from this chemotherapy AND
* For prior single administration of capecitabine: at least 6 months has elapsed between last capecitabine treatment and initiation of study treatment.
* For prior capecitabine-based combination regimen: at least 12 months has elapsed between last capecitabine-based treatment and initiation of study treatment.
* At least one unidimensionally measurable lesion according to RECIST criteria version 1.1.
* An Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2.
* Life expectancy of >3 months.
* Patients who are willing to undergo (oral) chemotherapy for the treatment of their disease and who are expected to comply with the treatment and study procedures, as per the Investigator's judgment.
* For women of child bearing potential, documented negative pregnancy test and agreement to use acceptable birth control measures during the duration of the study.
* Signed Informed consent obtained prior to any study related procedures.

Exclusion criteria:

* Patients who are HER 2 positive.
* Patients with 3 or more lines of chemotherapy failure for metastatic triple negative breast cancer.
* In ER/PR positive breast cancer, recurrence of the disease following 2 or more lines of chemotherapy failure and/or 3 or more lines of hormonal therapy failure.
* Patients presenting with de novo stage IV metastatic breast cancer, not previously treated for their disease.
* Patients who have already received any metronomic chemotherapy regimen.
* Known hypersensitivity to capecitabine or to any of its components.
* Known hypersensitivity to 5-fluorouracil.
* Known hypersensitivity to cyclophosphamide or any of its components.
* History of bladder carcinoma.
* Systemic anticancer therapy (chemotherapy, hormone therapy, or radiotherapy) within 4 weeks of randomization for the study.
* History of unexplained hematuria.
* History of dihydropyrimidine dehydrogenase (DPD) deficiency.
* Severe renal impairment (creatinine clearance below 30 mL/min [Cockroft and Gault]).
* Concomitant warfarin treatment.
* History of significant cardiac disease (eg, unstable angina, congestive heart failure, myocardial infarction, ventricular arrhythmias) within the previous 6 months.
* Conditions/situations such as:
* Patient is the Investigator or any Sub-Investigator, research assistant, pharmacist, Study coordinator, other staff, or relative thereof, directly involved in the conduct of the protocol.
* Uncooperative Patient or any condition that could make the Patient potentially noncompliant to the study procedures.
* Pregnant or breast-feeding women.
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Patients with a possibility of active tuberculosis as suggested by:
* Any signs or symptoms suggestive of active tuberculosis upon medical history or clinical examination.
* Chest radiograph within 3 months prior to the screening visit consistent with tuberculosis infection.
* Patients with close contact with a person with active tuberculosis.
* Known history of Human Immunodeficiency Virus (HIV).
* Any other significant medical conditions which in the judgment of the Investigator would preclude completion of the study.
* Participation in a clinical research study evaluating another investigational drug or therapy within 30 days prior to the Screening Visit.
* Presence of any of the following laboratory abnormalities at the Screening Visit:
* Hemoglobin <8.5 g/L;
* White blood cell (WBC) <3000/μL;
* Platelet count <100 000/μL;
* Absolute neutrophil count (ANC) <1500/μL;
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN) (or > 5 x ULN in patients with liver metastasis);
* Total Bilirubin >1.5 X ULN (or > 2 x ULN in patients with liver metastasis).
* Patients with a body surface area (BSA) <1.0 m² or 1.8 m².

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-01-23 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adverse events | 12 weeks
Assessment of PK parameter: maximum concentration (Cmax) | Daily 12 weeks
Assessment of PK parameter: time to reach Cmax (Tmax) | Daily 12 weeks

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 12 weeks
Objective Response Rate (ORR) | 12 weeks
Time to Progression (TTP) | 12 weeks
Proportion of patients compliant with treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- India (5):
  - Investigational Site Number 356009, Kollkata
  - Investigational Site Number 356002, Mumbai
  - Investigational Site Number 356007, New Delhi
  - Investigational Site Number 356008, Trivandrum
  - Investigational Site Number 356001, Vellore